CLINICAL TRIAL: NCT00889434
Title: Single-site, Open-label, Dose-ranging, Efficacy, and Safety Study of EGCG/Tocotrienol in 18 Patients With Splicing-mutation-mediated CF
Brief Title: Efficacy and Safety Study of EGCG/Tocotrienol in 18 Patients With Splicing-mutation-mediated Cystic Fibrosis (CF)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ECGC-TOC-HMO-CTIL
Record Dates: First submitted 2009-04-20; First posted 2009-04-28 (Estimated); Last update posted 2017-11-30 (Actual); Status verified 2017-02

CONDITIONS: Cystic Fibrosis
Keywords: Cystic fibrosis; splicing mutations; molecular therapy; EGCG; Tocotrienol; Splicing-mutation-mediated Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Tocotrienols; epigallocatechin gallate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- EGCG (Active Comparator): Two cycles comprising 28 days of continuous daily treatment with EGCGgiven 2 times/6 soft gel capsules (total 600 mg) /day (BID) in the morning and in the evening with food followed by a 14 day wash out period without drug.
  Interventions: Dietary Supplement: ECGC
- Tocotrienol (Active Comparator)
  Interventions: Dietary Supplement: Tocotrienol
- EGCG + Tocotrienol (Other): Combination of both arms
  Interventions: Dietary Supplement: EGCG + Tocotrienol

INTERVENTIONS:
Dietary Supplement: ECGC — 1 cycle will comprise 28 days of continuous daily treatment with EGCG given once/day(total 375 mg) /day in the morning with food followed by a 14 day wash out period without drug.
  Arms: EGCG
Dietary Supplement: Tocotrienol — One cycle will comprise 28 days of continuous daily treatment with Tocotrienol given 2 times/6 soft gel capsules (total 600 mg) /day (BID) in the morning and in the evening with food followed by a 14 day wash out period without drug.
  Arms: Tocotrienol
Dietary Supplement: EGCG + Tocotrienol — combination of both arms 375 mg EGCG + 600mg/day Tocotrienol
  Arms: EGCG + Tocotrienol

SUMMARY:
* Working Hypothesis: EGCG and Tocotrienol can act as genetic modifiers and increase the level of correctly spliced CFTR transcripts.
* Aims of the Study: To determine in patients with CF if oral administration of EGCG and Tocotrienol, both separate and in combination, modify CFTR splicing towards normal splicing as evaluated by improved Transepithelial Potential Difference (TEPD) assessment of chloride secretion.

To assess the effect of EGCG and Tocotrienol, both separate and in combination, on (1) additional TEPD measures of ion channel activity, (2) levels of correctly spliced CFTR mRNA in nasal mucosa, (3) cytokine levels in sputum and (4) changes in pulmonary function over the course of the study.

* Potential Implications to Medicine: Alternative splicing mechanisms are a common cause of genetic disease as ~15% of all known human mutations result in defective pre-mRNA splicing. Therapies based on augmenting the levels of full length or fully functioning proteins may have a substantial impact on the treatment of patients with genetic diseases.
* Contribution of the expected outcome to society Today genetic diseases can be treated but not healed. This proposal may be a step in the direction of finding a cure for patients carrying splicing mutations.

DETAILED DESCRIPTION:
Background: Cystic fibrosis (CF) is an autosomal recessive disorder caused by mutations in the CF trans-membrane conductance regulator protein. Despite substantial progress achieved in the understanding of the molecular basis and physiopathology of CF, a cure is not available. Mutation specific therapy is a novel approach to overcome the molecular defect in CF. We have previously shown that gentamicin and PTC 124 can induce read-through of nonsense CFTR mutations, and lead to functional CFTR. In addition we have shown that in vitro treatment with (-)epigallocatechin gallate (EGCG) and or Tocotrienol of cells harboring splicing mutations can augment production of full-length transcripts of affected proteins.

Working hypothesis and aims: EGCG and tocotrienol can act as genetic modifiers and increase the level of correctly spliced CFTR transcripts. Aim: To determine in CF patients if oral administration of EGCG and/or Tocotrienol, will modify CFTR splicing, as assessed by (1) Transepithelial Potential Difference (TEPD) as a measurement of ion channel activity, (2) levels of correctly spliced CFTR mRNA in nasal mucosa, (3) cytokine levels in sputum and (4) pulmonary function (FEV1).

Methods: Patients with CF carrying splicing mutations will be treated with EGCG 200 mg/day, Tocotrienol 600mg/day or both for 28 day cycles. Clinical parameters (TEPD, FEV1 and cytokine levels in sputum) and molecular parameters (mRNA levels,) will be analyzed to determine the effectiveness of the treatment.

Expected results: In vitro studies with cell cultures derived from CF patients have shown positive results; therefore an improvement in TEPD will be an indication for CFTR expression. An increase in mRNA levels and changes in FEV1, and cytokine levels will confirm the results.

Importance: Genetic therapy has encountered many technical difficulties. It is therefore of importance to develop alternative molecular strategies that will lead to an improvement or to a cure of genetic diseases.

Probable implications to Medicine: Alternative splicing mechanisms are a common cause of genetic disease as ~15% of all known human mutations result in defective pre-mRNA splicing. Therapies based on augmenting the levels of full length or fully functioning proteins may have a substantial impact on the treatment of patients with genetic diseases.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of CF.
2. Abnormal chloride secretion as measured by TEPD (a less than -5 mV TEPD assessment of chloride secretion with chloride-free amiloride and isoproterenol).
3. Presence of a splicing mutation in at least one allele of the CFTR gene.
4. Willingness and ability to comply with scheduled visits, drug administration plan, study procedures (including TEPD measurements, clinical laboratory tests,), and study restrictions.
5. Ability to provide written informed consent.
6. Evidence of personally signed and dated informed consent document indicating that the patient has been informed of all pertinent aspects of the trial.

Exclusion Criteria:

1. Prior or ongoing medical condition (e.g., concomitant illness, alcoholism, drug abuse, psychiatric condition), medical history, physical findings, ECG findings, or laboratory abnormality that, in the investigator's opinion, could adversely affect the safety of the patient, makes it unlikely that the course of treatment or follow-up would be completed, or could impair the assessment of study results.
2. Ongoing acute illness including acute upper or lower respiratory infections within 2 weeks before start of study treatment.
3. History of major complications of lung disease (including recent massive hemoptysis or pneumothorax) within 2 months prior to start of study treatment.
4. Abnormalities on screening chest x-ray suggesting clinically significant active pulmonary disease other than CF, or new, significant abnormalities such as atelectasis or pleural effusion which may be indicative of clinically significant active pulmonary involvement secondary to CF.
5. Abnormal liver function (serum ALT, AST, GGT, alkaline phosphatase, LDH, or total bilirubin > 2 times upper limit of normal). Abnormal renal function (serum creatinine >1.5 times upper limit of normal).
6. Pregnancy or breast-feeding.
7. History of solid organ or hematological transplantation.
8. Ongoing participation in any other therapeutic clinical trial or exposure to another investigational drug within 14 days prior to start of study treatment.
9. Change in intranasal medications (including use of corticosteroids, cromolyn, ipratropium bromide, phenylephrine, or oxymetazoline) within 14 days prior to start of study treatment.
10. Change in treatment with systemic or inhaled corticosteroids within 14 days prior to start of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2011-11-01 (Actual); Primary Completion 2015-04-16 (Actual); Study Completion 2015-04-16 (Actual)

PRIMARY OUTCOMES:
Changes in nasal chloride secretion as assessed by TEPD, with assessment of mean changes in TEPD by drug compared to baseline and the proportion of patients with a chloride secretion response by drug compared to baseline | 3 months

SECONDARY OUTCOMES:
Pulmonary function testing: forced expiratory volume in 1 sec [FEV1], forced vital capacity [FVC], and maximal expiratory flow25-75 [MEF25-75] | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Eitan Kerem, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Mount Scopus, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No